CLINICAL TRIAL: NCT06374511
Title: The Complications and Outcomes of Acutely Decompensated Cirrhosis: a Multi-center Nested Cohort Study
Brief Title: Prospective Cohort Study of Complications and Outcomes in Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-546
Record Dates: First submitted 2024-04-07; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Decompensated Cirrhosis; CMV Reactivation; Overt Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat from whole blood, urine samples, stool samples and peripheral blood mononuclear cell
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Inpatients diagnosed with decompensated cirrhosis form the Hepatology Unit, Nanfang Hospital, China. All patients with clinically verified diagnosis, irrespective of disease stage and etiology is included.
  Interventions: Diagnostic Test: Test for CMV reactivation

INTERVENTIONS:
Diagnostic Test: Test for CMV reactivation — All enrolled patients are monitored for CMV reactivation and hepatic encephalopathy using regular clinical tests or library test
  Other Names: Test and examine the severity of hepatic encephalopathy

SUMMARY:
This is a multi-center, nested cohort study intended to investigate the prevalence, risk factors, and outcomes of complications in patients with acutely decompensated cirrhosis, especially focused on Cytomegalovirus (CMV) reactivation, bacterial infections, hepatic encephalopathy, and Hepatorenal syndrome. Patients diagnosed with acutely decompensated cirrhosis were enrolled. Upon enrollment, detailed baseline data were collected and samples were harvested. Complications were assessed during hospitalization. Post-discharge follow-up was conducted through telephonic interviews at Day 30 and Day 90.

DETAILED DESCRIPTION:
This is a multi-center, nested cohort study intended to investigate the prevalence, risk factors, and outcomes of complications in patients with acutely decompensated cirrhosis, especially focused on CMV reactivation, bacterial infections, hepatic encephalopathy, and Hepatorenal syndrome. Patients diagnosed with acute decompensated cirrhosis were enrolled. Upon enrollment, detailed baseline data were collected and samples including ascites, feces, plasma, urine and PBMC were harvested. Following enrollment, patients were subjected to a rigorous follow-up regimen extending over a period of 90 days. Complications were assessed every 3-4 days during hospitalization through a combination of laboratory and clinical evaluations. Post-discharge follow-up was conducted through telephonic interviews at Day 30 and Day 90. Upon the emergence of new complications, such as infections (viral, bacterial or fungal) or hepatic encephalopathy, a detailed, complication-specific protocol was activated (Per complications protocols as follows).

Special complications protocols:

Hepatic encephalopathy:

1. The feces, plasma, and urine were collected at hepatic encephalopathy diagnosis before treatment and at Day 4, 7, 14 since hepatic encephalopathy treatment. If patients were discharged before14 days post-hepatic encephalopathy, the sample at discharge were collocated;
2. The treatment strategy for HE is recorded;
3. The HE severity assessments were carried out daily.

CMV reactivation:

1. The patients' plasma were collected twice a week for the assessment of CMV reactivation; The patients' peripheral blood mononuclear cells (PBMC) samples were collected at baseline and at the time of diagnosis of CMV reactivation;
2. The treatment strategy for CMV is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent
* Age between 18 years and 80 years
* Cirrhosis based on liver histology or a combination of characteristic clinical, biochemical, and imaging features
* Complications of decompensated cirrhosis (ascites, gastrointestinal bleeding and hepatic encephalopathy)

Exclusion Criteria:

* Malignancy
* Acquired immune deficiency syndrome
* Received immunosuppressive drugs for non-hepatic reasons
* Received organ transplantations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with liver cirrhosis, irrespective of time and circumstances of diagnosis, comorbidities and severity of disease will be offered inclusion in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of CMV reactivation | From enrollment to 90 days
  Cytomegalovirus DNA was quantified in stored plasma samples using real-time PCR (polymerase chain reaction) assay. DNA extraction was performed on 200 µL of plasma using a QIAamp DNA blood kit (Qiagen, German). Then, 25 µL of Tris (10 mM, pH 8.0) was used to elute the DNA, and 10 µL of the DNA was used for each PCR reaction. The minimum detection level was 102 copies/ml of plasma and values over this lower detection limit were considered to be CMV reactivation positive.
Incidence of hepatic encephalopathy | From enrollment to 90 days
  Patients meet West Haven criteria (Grade 1-4) were diagnosed of hepatic encephalopathy.

SECONDARY OUTCOMES:
Response to anti-CMV therapy | From CMV reactivation to one week and 90 days after treatment
  Patients with CMV reactivation may receive anti-CMV therapy; response to anti-CMV therapy was defined as patients' CMV-DNA test negative at more than 2 times.
Response to treatment for hepatic encephalopathy (HE) | From HE diagnosis to one week and 90 days after treatment
  Patients with hepatic encephalopathy may receive lactulose and (or) rifaximin; Patients' extent of HE change to Grade 0 (West Haven criteria) or decreased 2 grade from the baseline were be defined to response to the HE treatment.
Survival | From enrollment to 90 days
  Transplantation free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China